CLINICAL TRIAL: NCT03027596
Title: Remote Ischemic Conditioning to Reduce Burn Wound Progression
Acronym: RIC in burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BG Trauma Center Tuebingen (Other)
Responsible Party: Principal Investigator, Jens Rothenberger, Dr.med, BG Trauma Center Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 639/2016
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic conditioning (Experimental): Four cycles of 5 min occlusion and reperfusion in an extremity using a tourniquet.
  Interventions: Procedure: Remote ischemic conditioning
- Control group (No Intervention): no intervention

INTERVENTIONS:
Procedure: Remote ischemic conditioning
  Arms: Remote ischemic conditioning

SUMMARY:
Burned skin areas, which were initially vital, can be irreversibly damaged by wound progression. The aim of the present study is to evaluate the feasibility of ischemic conditioning to reduce secondary wound progression.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the study information and the consent to sign

  * Thermal injury (burn / scalding) with a clinical evaluated depth of at least 2a (superficial partial)
  * At least one of the following sites must not have skin lesions

    : Upper arm right and left
  * hospital admission within 6 hours after trauma has taken place

Exclusion Criteria:

* Participation in another experimental study

  * Pregnancy (women are subjected to a pregnancy test (urine)
  * Contraindication for the use of the tourniquet, for example Lymph drainage disorders after axillary lymphadenectomy or Irradiation of the axilla
  * Non-compliant patients who are, e.g. Intubated
  * Pure 3rd degree burns (full thickness) or charring
  * Thermal injuries older than 6 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change of burn depth | day 0, 1, 2, 3, 4,5, 7, 11,18,21, 90,180
  Clinical assessment of burn depth

SECONDARY OUTCOMES:
Change in skin's relative amount of hemoglobin | day 0, 1, 2, 3, 4,5, 7, 11,18,21, 90,180
  relative amount of hemoglobin (Arbitrary Units)
Change in skin's blood flow | day 0, 1, 2, 3, 4,5, 7, 11,18,21, 90,180
  blood flow (Arbitrary Units)
Change in skin's oxygen saturation | day 0, 1, 2, 3, 4,5, 7, 11,18,21, 90,180
  oxygen saturation (%)
Change in skin elasticity | day 0, 1, 2, 3, 4,5, 7, 11,18,21, 90,180, 360
  objective measurement of the skin elasticity
Differences in scare development between the study groups | day 90, 180, 360
  Assessment with the Vancouver scare scale

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rothenberger, M.D., Principal Investigator — Hand and Plastic Surgery, BG Trauma Center Tübingen, Germany
Locations (1):
- BG Trauma Center, University Tübingen, Germany, Tübingen, Germany, Germany

IPD SHARING:
Plan to Share IPD: Undecided